CLINICAL TRIAL: NCT01419782
Title: The Effects Of Femur On The Resting Myoelectrical Activity Of Contralateral Adductor Muscle During Unilateral Lower Extremity Vibration: Bone Myoregulation Reflex
Brief Title: Effects of Unilateral WBV on Muscleactivity of Contralateral Hip Adductor
Acronym: WBV-BM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ilhan Karacan, Clinical Associated Professor, ILHAN KARACAN, Bagcilar Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: BEAH FTR-5
Record Dates: First submitted 2011-08-17; First posted 2011-08-18 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Bone Mass; Effects of Vibration
Keywords: bone; osteocyte; rest muscle electrical activity; whole-body vibration; sclerostin
MeSH Terms: conditions — Sclerosteosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Whole-body vibration (Experimental): whole body vibration will be applied the right lower limb.
  Interventions: Other: Whole-body vibration

INTERVENTIONS:
Other: Whole-body vibration — Frequency: 40 Hz, vibration amplitude: 2 mm, duration: 60 sec
  Other Names: Cyclic mechanical loading

SUMMARY:
The aim of this study is to investigate effects of femur exposed to unilateral vibration on the rest muscle electrical activity of contralateral hip adductors and contralateral soleus H-reflex in young adult men.

This study hypothesize that femur exposed to unilateral vibration may affect the rest muscle electrical activity of contralateral hip adductors. Vibration can effectively enhance muscle strength and power. Previous studies have shown that vibration increases muscle electromyographic (EMG) activity. It has been showed that bone has an effect on the increase in muscle EMG activity caused by vibration in healthy young adults in a study. In this study, it was reported that vibrations-induced increases in muscle electrical activity of flexor carpi radialis (FCR) was related to ultradistal radius bone mineral content (BMC) and the FCR H-reflex was suppressed or depressed during vibration. This findings were reported to support the assumption that the bone exposed to cyclic mechanical loading may neuronally regulate muscle activity.

DETAILED DESCRIPTION:
A total of 20 voluntaries are planned to include in this study.

Vibration will be applied the right lower extremity by whole-body vibration (PowerPlate Pro). Cases will stand on vibration plate. WBV will be applied at a frequency of 40 Hz and amplitude of 2 mm for 60 seconds. WBV will be applied one session only.

The rest muscle electrical activity of ipsilateral and contralateral hip adductor muscles at rest will be measured by PowerLab (data acquisition system, ADInstruments, Australia) device.The rest-EMGrms will be measured at before and during vibration. We also evaluate a change in contralateral soleus H reflex during vibration.

Effects of bone on the rest muscle electrical activity will be assessed by hip bone mineral density, bone mineral content and serum sclerostin level. The right hip bone mineral density (BMD) and BMC will be evaluated by bone densitometer (Norland). Plasma sclerostin level will be measured by using Human Sclerostin ELISA kıt before and after vibration.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-40 yrs
* Gender: Male
* Volunteer
* Healthy status: Patients having hypoesthesia in his leg and Healthy subjects
* Dominant hand:Right-handed

Exclusion Criteria:

* Bone diseases (osteoporosis, osteomalacia, paget's disease, neoplasm, etc),
* Systemic diseases (cardiovascular, endocrine, infections etc),
* Myopathy-tendinopathy
* Lower limb joint disease
* Vertigo
* Obesity (BMI >30 kg/m2)
* Professional sportsman
* Male doing regular sports activities
* Skin disease in lower limb
* Non-cooperative subject
* Hemolysis of blood sample

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-03; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Vibration-induced contralateral muscle electrical activity | 3 month

CONTACTS AND LOCATIONS:
Overall Officials: ILHAN KARACAN, MD, Principal Investigator — Bagcilar Training & Research Hospital
Locations (1):
- Bagcilar Training & Research Hospital, Istanbul, Turkey (Türkiye)